CLINICAL TRIAL: NCT01097226
Title: Bioavailability and Vascular Effects of Apple Polyphenols
Acronym: POLYMALUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Danisco (Industry); Coressence LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IFR06-2009
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Dietary intervention; bioavailability; Healthy volunteers
MeSH Terms: interventions — Catechin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apple flavanols (Experimental)
  Interventions: Other: Apple extract delivering 70 mg epicatechin; Other: Apple extract delivering 140 mg epicatechin; Other: Apple granules delivering 70 mg epicatechin; Other: Water delivering no epicatechin

INTERVENTIONS:
Other: Apple extract delivering 70 mg epicatechin — Delivered as a flavoured water based beverage
Other: Apple extract delivering 140 mg epicatechin — Delivered as a flavoured water based beverage
Other: Apple granules delivering 70 mg epicatechin — Delivered as a puree
Other: Water delivering no epicatechin — Delivered as flavoured water

SUMMARY:
The main purpose of this study is to determine the oral bioavailability of flavanols (polyphenolic compounds) from apple granules and an apple extract delivered in a water based beverage at two different doses. We will also investigate the effects of apple flavanols on nitric oxide production.

DETAILED DESCRIPTION:
This study is a randomized four phase crossover trial investigating the bioavailability of apple flavanols and the effects on nitric oxide products, a surrogate marker for changes in endothelial function. Each test phase will comprise a 3 day period of intervention which will be identical in nature (except for the test product consumed) and separated by a minimum of 1 week. On days 1-3 of each test phase volunteers will consume a low flavanol diet. After consumption of the test product on the morning of day 2, blood and urine samples will be collected at regular intervals for the next 24h.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 45-70 years

Exclusion Criteria:

* Smokers (or have quit smoking less than 1 year ago)
* Regular prescribed medication (excluding some eye and skin medication that is judged not to affect study outcome)
* Non-prescribed medication that may affect the study data, e.g. aspirin. The use of non prescribed medications will be assessed on an individual basis.
* Dietary supplements or herbal remedies which may affect the study data unless the volunteer is willing to discontinue them for 1 month prior to starting study. (Please note that some supplements may not affect the study and this will be assessed on an individual basis).
* Gastro-intestinal diseases (excluding hiatus hernia unless symptomatic or study intervention/procedure is contra-indicated).
* Diabetics
* Known cardiovascular disease
* Asthmatics (unless no medication taken for 1 year)
* Lactose Intolerance
* Pregnancy or have been pregnant within the last 12 months
* Parallel participation in another research project which involves dietary intervention
* Participation in another research project which has involved blood sampling within the last four months unless the total amount of combined blood from both studies does not exceed 470 mls.
* Has donated or intends to donate blood within 16 weeks prior to or during the study period.
* Depressed or elevated blood pressure measurements (<90/50 or 95/55 if symptomatic or >160/100)
* Any person related to or living with any member of the study team
* Results of the clinical screening which indicate or are judged by the HNU Medical Advisor to be indicative of a health problem which could compromise the well-being of the volunteer if they participated or which could affect the study data.
* Alcohol consumption > approximately 20 g alcohol/day (2.5 units/day)
* BMI <19.5 or > 35

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma pharmacokinetic curve for total epicatechin | 24 hours

SECONDARY OUTCOMES:
Additional measures of bioavailability: Plasma Cmax, Tmax, half life and urinary excretion | 24 hours
Changes in levels of nitric Oxide metabolites as a surrogate measure of endothelial function after consumption of apple flavanols | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kroon, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Saha S, Hollands W, Needs PW, Ostertag LM, de Roos B, Duthie GG, Kroon PA. Human O-sulfated metabolites of (-)-epicatechin and methyl-(-)-epicatechin are poor substrates for commercial aryl-sulfatases: implications for studies concerned with quantifying epicatechin bioavailability. Pharmacol Res. 2012 Jun;65(6):592-602. doi: 10.1016/j.phrs.2012.02.005. Epub 2012 Feb 25. PMID 22373658